CLINICAL TRIAL: NCT04025788
Title: BIOTRONIKS-Safety and Performance in de Novo Lesion of Native Coronary Arteries With Magmaris (BIOSOLVE)-IV Magmaris Swiss Satellite Registry
Brief Title: BIOSOLVE-IV Magmaris Swiss Satellite Registry
Status: Terminated | Type: Observational
Why Stopped: Slow enrolment. New generation BRS available
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, IGLESIAS Juan Fernando, Medical Doctor, Principal Investigator, University Hospital, Geneva
Other Study IDs: 2018-01420
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Magmaris Resorbable Magnesium Scaffold (RMS) — Subjects will undergo a percutaneous coronary intervention for the implantation of the Magmaris scaffold in accordance with the standard of care and standard hospital practice. Maximum of two single de novo lesions in two separate major epicardial vessels are allowed.

SUMMARY:
BIOSOLVE-IV Magmaris Swiss Satellite Registry is a prospective, single-arm, multicenter, nationwide open label registry. It is planned to enroll 200 subjects in up to 12 participating sites in Switzerland. After percutaneous coronary intervention (PCI) with the Magmaris scaffold and signature of the informed consent form, all subjects will be followed through hospital discharge and will undergo follow up evaluations at 6, 12 and 24 months post procedure. The follow up evaluations, part of the standard care can be either performed on site (12 months) or by phone (6 and 24 months) and according to routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥18 years of age
* Subject must be willing to sign a Patient Informed Consent
* Symptomatic coronary artery disease
* Subject with a maximum of two single de novo lesions in two different major epicardial vessels
* Target lesion length ≤ 21 mm by QCA or by visual estimation
* Target lesion stenosis >50% and <100% by visual estimation, and TIMI flow ≥1.
* Subject is eligible for Dual Anti Platelet Therapy (DAPT)
* Reference vessel diameter between 2.7-3.7 mm by visual estimation, depending on the scaffold size used

Exclusion Criteria:

* Pregnant and/or breastfeeding females or females who intend to become pregnant during the time of the registry
* Known allergies to: Acetylsalicylic Acid (ASA), clopidogrel, heparin or any other anticoagulant /antiplatelet required for PCI, contrast medium, sirolimus, or similar drugs; or the scaffold materials including Magnesium, Yttrium, Neodymium, Zirconium, Gadolinium, Dysprosium, Tantalum that cannot be adequately pre-medicated
* Subjects on dialysis
* Subject has clinical symptoms and/or electrocardiogram (ECG) changes consistent with acute ST elevation myocardial infarction (STEMI) within 72 hours prior to the index procedure. Note: Hemodynamically stable non-STEMI (NSTEMI) subjects are eligible for study enrollment
* Documented left ventricular ejection fraction (LVEF) ≤30% as documented within maximum 6 months prior to the procedure
* Heavily calcified or extremely tortuous lesions
* Bifurcation lesion requiring side branch intervention, if side branches >2 mm in diameter are involved
* Restenotic target lesion
* Thrombus in target vessel
* Target lesion is located in or supplied by a diseased (defined as vessel irregularity per angiogram and >20% stenosed lesion by visual estimation) arterial or venous bypass graft
* Left main coronary artery disease
* Ostial target lesion (within 5.0 mm of vessel origin)
* Target vessel (including side branches) has second lesion which requires treatment according to the investigator's discretion
* Unsuccessful pre-dilatation, defined as residual stenosis rate >20% by visual estimation and/or angiographic complications (e.g. distal embolization, side branch closure, extensive dissections)
* Planned surgery within 6 months of PCI unless dual antiplatelet therapy will be maintained
* Currently participating in another study and primary endpoint is not reached yet
* Planned interventional treatment of any non-target vessel within 30 days post procedure
* Planned intervention of the target vessel within 6-month after the index procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: BIOSOLVE-IV Magmaris Swiss Satellite Registry will include male and female subjects requiring a treatment of de novo coronary artery lesions with Magmaris.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Target Lesion Failure at 12 months | 12 months
  Target Lesion Failure (TLF, a composite of cardiac death, target vessel Q-wave or non-Q wave Myocardial Infarction, and clinically driven Target Lesion Revascularization) at 12 months

SECONDARY OUTCOMES:
Target Lesion Failure | 6 months and annually thereafter up to 2 years post-procedure
  Target Lesion Failure (TLF) at 6, 12 and 24 months
Clinically driven Target Lesion Revascularization | 6, 12 months and 24 months post-procedure
  Clinically driven Target Lesion Revascularization (TLR) at 6, 12 and 24 months
Clinically driven Target Vessel Revascularization | 6, 12 months and 24 months post-procedure
  Clinically driven Target Vessel Revascularization (TVR) at 6, 12 and 24 months
Cardiac death | 6, 12 and 24 months post-procedure
  Cardiac death at 6, 12 and 24 months
Target Vessel Myocardial Infarction | 6, 12 and 24 months post-procedure
  Target Vessel Myocardial Infarction (MI) at 6, 12 and 24 months
Scaffold thrombosis | 6, 12 and 24 months post-procedure
  Scaffold thrombosis at 6, 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Juan F Iglesias, MD, Principal Investigator — University Hospital, Geneva
Locations (6):
- Switzerland (6):
  - Unité de Cardiologie interventionnelle, Service de cardiologie, Hôpitaux Universitaires de Genève, Geneva
  - Kantonsspital Baselland, Kardiologie, Liestal
  - Ensemble Hospitalier de la Côte, Hôpital de Morges, Cardiologie, Morges
  - Interventionnelle Kardiologie, Kantonspital St.Gallen, Kardiologie, Sankt Gallen
  - Hôpital du Valais Sion, Sion
  - HFR Fribourg, Cardiologie, Villars-sur-Glâne